CLINICAL TRIAL: NCT02812719
Title: Comparing the Efficacy and Safety of Combined Glycolic Acid and Salicylic Acid Peel Versus Glycolic Acid Peel Alone in the Treatment of Melasma: A Split Face Study
Brief Title: Treatment of Melasma With Glycolic Acid-Salicylic Acid Peel Versus Glycolic Acid Peel
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study did not receive funding and will not be implemented.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-33976
Record Dates: First submitted 2015-10-28; First posted 2016-06-24 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Glycolic acid peel alone (Active Comparator): One of two sides of the face will be randomly treated with glycolic acid peel 35% alone.
  This treatment will be administered at visit 1 (but to entire face) and 3 subsequent visits (to one randomly selected side of the face), for a total of 4 treatments at 2 week intervals
  Interventions: Drug: Glycolic acid peel alone
- Glycolic and salicylic acid peel (Experimental): The other randomly chosen side of the face will be treated with glycolic acid peel 35% followed by salicylic acid peel 20%, as a combination treatment.
  This treatment will be administered at visits 2, 3 and 4 (to one randomly selected side of the face), for a total of 3 treatments at 2 week intervals.
  Interventions: Drug: Glycolic and salicylic acid peel

INTERVENTIONS:
Drug: Glycolic acid peel alone — One of two sides of the face will be randomly treated with glycolic acid peel 35% alone.
  This treatment will be administered at visit 1 (but to entire face) and 3 subsequent visits (to one randomly selected side of the face), for a total of 4 treatments at 2 week intervals
  Other Names: Single acid skin peel
  Arms: Glycolic acid peel alone
Drug: Glycolic and salicylic acid peel — The other randomly chosen side of the face will be treated with glycolic acid peel 35% followed by salicylic acid peel 20%, as a combination treatment.
  This treatment will be administered at visits 2, 3 and 4 (to one randomly selected side of the face), for a total of 3 treatments at 2 week intervals.
  Other Names: Combination acid skin peel
  Arms: Glycolic and salicylic acid peel

SUMMARY:
The aim of this pilot study is to conduct a controlled comparison of the efficacy and safety of a combination peel (glycolic acid and salicylic acid) as compared to glycolic acid peel alone in the treatment of melasma. Our primary outcome is objective improvement in pigmentation as evaluated using a colorimeter. Our secondary outcomes are subjective improvement using the Melasma Area and Severity Index (MASI) and Patient and Physician Global assessment, as well as assessment of treatment tolerability and patient satisfaction.

DETAILED DESCRIPTION:
Melasma is an acquired form of hyperpigmentation that is seen most commonly on the face, characterized by symmetrically distributed brown patches of variable darkness. The cosmetically unattractive nature of this disorder has been shown to negatively affect a patient's quality of life. Unfortunately, the treatment of melasma is challenging and often disappointing. Treatment includes a combination approach with strict sun protection, cosmetic camouflage, topical lightening agents, laser therapy, and chemical peels.

Today, the investigators define chemical peeling as the application of chemical exfoliating agents to the skin, which results in destruction of one or more parts of the epidermis and/or dermis with subsequent regrowth of these layers. Chemical peels are divided into superficial (light), medium, and deep; with superficial peels being the focus of this study. Superficial peels penetrate into the epidermis only, and are a safe, widely available and well-tolerated treatment modality. These peeling agents include glycolic acid, lactic acid, mandelic acid, salicylic acid and trichloroacetic acid, each with unique properties. For instance, alpha-hydroxy acids, such as glycolic acid, are known to be hydrophilic, whereas salicylic acid is lipophilic and anti-inflammatory.

As each peeling agent has unique properties, it can be hypothesized that the combined use of these agents may result in better clinical outcomes than the use of an agent alone. Prior studies have demonstrated that the combined use of these peels are safe and effective in improving a variety of skin conditions including acne scars, hyperpigmentation, and infraorbital dark circles. Overall however, studies on the combined use of these chemical peels in the treatment of melasma are lacking.

Therefore, the aim of this pilot study is to conduct a controlled comparison of the efficacy and safety of a combination peel (glycolic acid and salicylic acid) as compared to glycolic acid peel alone in the treatment of melasma.

ELIGIBILITY:
Inclusion Criteria:

* Female and males aged 18 or older
* Subjects with melasma on both sides of the face (forehead or cheek).
* Subjects in general good health
* Female of childbearing age will be on a reliable form of contraception during the course of treatment other than oral contraceptive pills or hormonal intrauterine device.
* Subjects must be willing to sign consent, answer questionnaires, comply with all clinical visits, and use sunscreen and sun-protection.
* Subjects must be willing to not apply other treatment options for melasma during the course of the study

Exclusion Criteria:

* Subjects suffering from other pigmentation disorders.
* Subjects with known allergy to any components of the peels
* Subjects who have active uncontrolled disease to facial area (i.e acne).
* Pregnant women, nursing mothers.
* Subjects with history of abnormal scaring
* Subjects who cannot communicate with investigators or who are unlikely to cooperate.
* Subjects in a situation in which in the opinion of the investigators, may interfere with optimal participation in the study.
* Subjects who have used chemical peels, microdermabrasion or facial laser treatments in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in pigmentation | Week 0, Week 7-8 (1-2 weeks following 4th peel), and Week 18 (12 weeks following 4th peel)
  Change in pigmentation using a colorimeter

SECONDARY OUTCOMES:
Change in pigmentation score | Week 0, Week 7-8 (1-2 weeks following 4th peel), and Week 18 (12 weeks following 4th peel)
  Change in pigmentation using the Melasma Area and Severity Index (MASI)
Improvement of melasma | Week 0 and Week 7-8 (1-2 weeks following 4th peel), and Week 18 (12 weeks following 4th peel)
  Improvement of melasma based on Patient and Physician Global assessment
Adverse events assessment | Week 7-8 (1-2 weeks following 4th peel)
  Patient questionnaire to assess for any adverse events encountered

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dominguez AR, Balkrishnan R, Ellzey AR, Pandya AG. Melasma in Latina patients: cross-cultural adaptation and validation of a quality-of-life questionnaire in Spanish language. J Am Acad Dermatol. 2006 Jul;55(1):59-66. doi: 10.1016/j.jaad.2006.01.049. Epub 2006 May 2. PMID 16781293
- [Background] Berson DS, Cohen JL, Rendon MI, Roberts WE, Starker I, Wang B. Clinical role and application of superficial chemical peels in today's practice. J Drugs Dermatol. 2009 Sep;8(9):803-11. PMID 19746672
- [Background] Kodali S, Guevara IL, Carrigan CR, Daulat S, Blanco G, Boker A, Hynan LS, Pandya AG. A prospective, randomized, split-face, controlled trial of salicylic acid peels in the treatment of melasma in Latin American women. J Am Acad Dermatol. 2010 Dec;63(6):1030-5. doi: 10.1016/j.jaad.2009.12.027. PMID 20889235
- [Background] Sarkar R, Kaur C, Bhalla M, Kanwar AJ. The combination of glycolic acid peels with a topical regimen in the treatment of melasma in dark-skinned patients: a comparative study. Dermatol Surg. 2002 Sep;28(9):828-32; discussion 832. doi: 10.1046/j.1524-4725.2002.02034.x. PMID 12269877
- [Background] Soliman MM, Ramadan SA, Bassiouny DA, Abdelmalek M. Combined trichloroacetic acid peel and topical ascorbic acid versus trichloroacetic acid peel alone in the treatment of melasma: a comparative study. J Cosmet Dermatol. 2007 Jun;6(2):89-94. doi: 10.1111/j.1473-2165.2007.00302.x. PMID 17524124
- [Background] Grimes PE. The safety and efficacy of salicylic acid chemical peels in darker racial-ethnic groups. Dermatol Surg. 1999 Jan;25(1):18-22. doi: 10.1046/j.1524-4725.1999.08145.x. PMID 9935087
- [Background] Lee HS, Kim IH. Salicylic acid peels for the treatment of acne vulgaris in Asian patients. Dermatol Surg. 2003 Dec;29(12):1196-9; discussion 1199. doi: 10.1111/j.1524-4725.2003.29384.x. PMID 14725662